CLINICAL TRIAL: NCT01083537
Title: Phase I/II Trial of Best Supportive Care and Chemotherapy, Either Cisplatin or Paclitaxel, in Patients With Primary Ovarian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer Presenting With Inoperable Malignant Bowel Obstruction
Brief Title: Trial of Best Supportive Care and Either Cisplatin or Paclitaxel to Treat Patients With Primary Ovarian Cancer, Primary Peritoneal Cancer or Fallopian Tube Cancer and Inoperable Malignant Bowel Obstruction
Status: Terminated | Phase: Phase 1 / Phase 2 | Type: Interventional
Why Stopped: Slow accrual
Sponsor: University Health Network, Toronto (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MBO-CHEMO-BSC
Record Dates: First submitted 2010-03-01; First posted 2010-03-09 (Estimated); Last update posted 2019-02-15 (Actual); Status verified 2019-02

CONDITIONS: Ovarian Cancer; Peritoneal Cancer; Fallopian Tube Cancer; Bowel Obstruction
Keywords: malignant bowel obstruction; ovarian cancer; Peritoneal cancer; Fallopian Tube cancer
MeSH Terms: conditions — Ovarian Neoplasms; Fallopian Tube Neoplasms; Intestinal Obstruction | interventions — Cisplatin; Paclitaxel

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Cisplatin (Experimental): Cisplatin administered at 60mg/m2 IV on Day 1, every 21 days for 2 cycles.
  1. Hesketh Level 5: 5HT3 receptor antagonist IV/po 30-60 mins pre-chemo and Dexamethasone 10-20mg po/IV 30-60 mins pre-chemo; Dexamethasone 4-8mg po BID x 3 days starting 24hours post last dose of chemo; Prochlorperazine 10mg po/IV q4-6h prn, metoclopramide 10-20mg po/iv q6h prn, haloperidol 0.5-2mg po/SC q 8-12 h prn
  2. Hydration: Pre-hydration 500-1000cc NS with 10Meq KCl over 2 hours; Infuse Cisplatin in 250-500cc NS over 1 hour; Post-hydration 1000cc NS + 20Meq KCl (+/- 2g MgSO4) over 1 hour
  Interventions: Drug: Cisplatin
- Paclitaxel (Experimental): Paclitaxel administered 80mg/m2 IV on Days 1, 8 and 15, every 21 days for 2 cycles.
  1. Suggested prophylaxis for paclitaxel-associated hypersensitivity reactions: Dexamethasone 10-20mg po/IV 30-60 mins pre-chemo; diphenydramine 25-50mg IV 30-60 minutes pre-chemo, ranitidine 50mg IV 30-60 minutes pre-chemo
  2. Hesketh Level 2: Prochlorperazine 10mg po/IV q4-6h prn
  3. Hydration: Infuse Paclitaxel in 250cc NS over 1 hour
  Interventions: Drug: Paclitaxel

INTERVENTIONS:
Drug: Cisplatin — 1) Cisplatin administered at 60mg/m2 IV on Day 1, every 21 days for 2 cycles.
  1. Hesketh Level 5: 5HT3 receptor antagonist IV/po 30-60 mins pre-chemo and Dexamethasone 10-20mg po/IV 30-60 mins pre-chemo; Dexamethasone 4-8mg po BID x 3 days starting 24hours post last dose of chemo; Prochlorperazine 10mg po/IV q4-6h prn, metoclopramide 10-20mg po/iv q6h prn, haloperidol 0.5-2mg po/SC q 8-12 h prn
  2. Hydration: Pre-hydration 500-1000cc NS with 10Meq KCl over 2 hours; Infuse Cisplatin in 250-500cc NS over 1 hour; Post-hydration 1000cc NS + 20Meq KCl (+/- 2g MgSO4) over 1 hour
  Arms: Cisplatin
Drug: Paclitaxel — 2) Paclitaxel administered 80mg/m2 IV on Days 1, 8 and 15, every 21 days for 2 cycles.
  1. Suggested prophylaxis for paclitaxel-associated hypersensitivity reactions: Dexamethasone 10-20mg po/IV 30-60 mins pre-chemo; diphenydramine 25-50mg IV 30-60 minutes pre-chemo, ranitidine 50mg IV 30-60 minutes pre-chemo
  2. Hesketh Level 2: Prochlorperazine 10mg po/IV q4-6h prn
  3. Hydration: Infuse Paclitaxel in 250cc NS over 1 hour
  Arms: Paclitaxel

SUMMARY:
The best way to treat MBO in patients with ovarian cancer has not been studied enough by trials that assess how more than one treatment arm (surgical, chemotherapeutic, supportive care approaches) affects clinical outcomes like resolution of bowel obstruction, survival, and quality of life. To improve patient outcomes, we must assess which patients will do better with palliative surgery, chemotherapy, or best supportive care. This study will gather safety information, and how reasonable it is to give chemotherapy and BSC to patients with advanced ovarian cancer and MBO who are non-surgical candidates. This study will also look into the effects of chemotherapy and BSC on the quality of life and resolution of bowel obstruction, in hopes to perform future studies that lead to the best management of MBO.

DETAILED DESCRIPTION:
The optimal management of MBO in patients with ovarian cancer has not been defined by proper prospective randomized control trials evaluating the impact of defined multidisciplinary treatment arms (surgical, chemotherapeutic, supportive care approaches) on important clinical outcomes including resolution of bowel obstruction, survival endpoints and validated quality of life outcomes. In order to improve patient outcomes, we must define which patients will benefit from palliative surgery, which patients are appropriate candidates for chemotherapy and which patients will benefit most from best supportive care. This study will determine the safety, feasibility of chemotherapy and BSC in patients with advanced ovarian cancer presenting with MBO who are initially deemed non-surgical candidates and will identify the impact of chemotherapy and BSC on quality of life and resolution of bowel obstruction, in preparation for future prospective randomized studies to determine the optimal management of MBO.

ELIGIBILITY:
Inclusion Criteria:

* Hospital admission and diagnosis compatible with Malignant Bowel Obstruction, as defined below:

  1. A diagnosis of primary ovarian cancer, primary peritoneal cancer or fallopian tube cancer
  2. At least two of the following four symptoms: (a) vomiting (>2 episodes in past 24 hours), (b) abdominal pain, (c) not passing gas per rectum in past 24 hours, (d) severe constipation (no bowel movement >24 hours).
  3. CT findings suggestive of complete bowel obstruction. CT Abdomen: confirms diagnosis of bowel obstruction (93% sensitivity 93-100% specificity) and aids in determining the location and etiology of obstruction.
* Non-surgical candidate
* Ability to understand and the willingness to sign a written informed consent document.
* Patients must be 18 years of age or older.
* ECOG performance status 0, 1 or 2 (Karnofsky > or = 60%) one week prior to admission.
* Patients must have adequate hematological function as defined below:
* Absolute granulocyte count > or = 1.5 x 10^9/L
* Platelet count > or = 100 x 10^9/L
* Patients must have adequate renal and hepatic function as defined below:
* Serum creatinine < or = 1.5 x ULN OR a calculated creatinine clearance > or = 50 ml/min
* Bilirubin < or = 3 x ULN, AST < or = 5 x ULN, ALT < or = 5 x ULN

Exclusion Criteria:

* Patients diagnosed with MBO caused by malignancy other than primary ovarian cancer.
* Patients diagnosed with MBO who are surgical candidates.
* Patients who are pregnant or breast-feeding.
* Concomitant diagnosis of GI malignancy (platinum ineffective) within past 5 years.
* History of severe hypersensitivity reaction to Cisplatin and Paclitaxel.
* Patients who have received chemotherapy within 2 weeks prior to study enrollment.
* Patients with uncontrolled Inflammatory Bowel Disease.
* Patients with concurrent active infections with Clostridium Difficile.
* Early postoperative obstruction (within 30 days from previous operation).
* Patients who have had bowel irradiation within 6 weeks.
* Patients with any of the following conditions are excluded:
* Myocardial infarction within 6 months prior to entry.
* Congestive heart failure.
* Unstable angina.
* Active cardiomyopathy.
* Unstable ventricular arrhythmia.
* Uncontrolled hypertension.
* Uncontrolled psychotic disorders.
* Serious infections.
* Active peptic ulcer disease.
* Uncontrolled psychiatric illness.
* Any other medical conditions that might be aggravated by treatment or limit compliance.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1 (Actual)
Dates: Start 2010-02; Primary Completion 2012-06 (Actual); Study Completion 2012-06 (Actual)

PRIMARY OUTCOMES:
Overall Safety Profile | Day 1 of treatment until resolution of symptoms
  Type, frequency, severity (NCI CTCAE v.3.0.1) and relationship to trial treatment of adverse events and laboratory abnormalities. Frequency and severity of adverse events will be tabulated using counts and proportions detailing frequently occurring, serious and severe events of interest.
Quality of Life Scores at Baseline, Day 30 and Day 90 | Day 1 of treatment until resolution of symptoms
  Quality of life scores will be tabulated using counts and summary statistics. We hypothesize that at 30 days from treatment, there may be no improvement in quality of life scores compared to baseline. We hypothesize that at 90 days from treatment, there will be an improvement in quality of life scores from baseline by one third standard deviation. Paired T test and Mixed model will be used to make the comparison over different time period.
Time to Resolution of Bowel Obstruction | Day 1 of treatment until resolution of symptoms
  Time to resolution of bowel obstruction and time to recurrence of bowel obstruction will be assessed using summary statistics including mean, median, counts and proportion, to summarize the patients.

SECONDARY OUTCOMES:
Survival | 30 days, 60 days, and 90 days from treatment start date
  Survival: 30-day(all cause and disease-specific), 60-day(all cause and disease-specific), and 90-day mortality (all cause and disease-specific).
  Summary statistics will be used to summarize the patients. Survival estimates will be computed using Kaplan-Meier method. Variable association will be measured using Pearson correlation coefficients, chi-square tests, one- or two-sample t-tests or logistic regression analyses. Non-parametric tests may be substituted if necessary. Results will be illustrated using figures and plots using 95 percent confidence intervals.
Evaluation of Toxicity | Time of consent until resolution of symptoms
  All patients will be evaluable for toxicity from the time they sign consent.

CONTACTS AND LOCATIONS:
Overall Officials: Amit Oza, Principal Investigator — Princess Margaret Hospital, Canada; Nicole Chau, Principal Investigator — Princess Margaret Hospital, Canada
Locations (1):
- Princess Margaret Hospital, Toronto, Ontario, Canada